CLINICAL TRIAL: NCT07279935
Title: Biomarker-Directed Treatment in Patients Who Had Distant Recurrence After Adjuvant Osimertinib for EGFRm Resectable SIB-IIIA NSCLC: A Prospective, Multi-cohort, Interventional Study (REVIVE)
Brief Title: Osimertinib Combined With Chemotherapy in Patients Who Had Distant Recurrence After Adjuvant Osimertinib for EGFRm Resectable SIB-IIIA NSCLC.
Acronym: REVIVE
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5164L00004
Record Dates: First submitted 2025-12-01; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases; Carcinoma, Non-Small-Cell Lung; osimertinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Bronchogenic; Bronchial Neoplasms; Lung Neoplasms; Respiratory Tract Neoplasms; Thoracic Neoplasms; Neoplasms by Site; Neoplasms; Lung Diseases; Respiratory Tract Diseases | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cohort1 (Experimental): Treatment allocation according to molecular profile at recurrence. Cohort 1 consists of patients with Ex19del or L858R mutation.
  Interventions: Drug: Osimertinib+cisplatin or carboplatin + pemetrexed Edit

INTERVENTIONS:
Drug: Osimertinib+cisplatin or carboplatin + pemetrexed Edit — Cohort 1 treated with osimertinib 80 mg once daily (QD) in combination with platinum-based chemotherapy cisplatin [75 mg/m2] or carboplatin [AUC5]) plus pemetrexed (500 mg/m2) on Day 1 every 3 weeks (Q3W) for 4 cycles, followed by osimertinib QD and pemetrexed Q3W till RECIST 1.1-defined progression or until another discontinuation criterion is met.
  Other Names: Cohort1

SUMMARY:
This study is designed as a multi-cohort trial based on various patient biomarkers study with the potential to include new study treatment in the future. EGFR-sensitive mutation-positive patients with distant recurrence after adjuvant osimertinib treatment for EGFRm resectable SIB-IIIA NSCLC and scheduled to receive osimertinib plus chemotherapy will be enrolled in cohort 1. In this cohort, approximately 100 patients will be recruited from 25 sites in China. The enrolment period is planned to be approximately 16 months.

ELIGIBILITY:
Inclusion Criteria for pre-screening:

1. Prior complete surgical resection (R0) and adjuvant osimertinib in EGFRm resectable SIB-IIIA NSCLC (AJCC 7th edition).
2. Off-treatment recurrence (including completed 3 years adjuvant osimertinib & discontinued adjuvant osimertinib before 3 years due to non-recurrence reason).
3. Newly diagnosed distant recurrent NSCLC (IVA or IVB) (per Version 9 of the International Association for the Study of Lung Cancer [IASLC] Staging Manual in Thoracic Oncology).
4. ≥6 months interval between recurrence and completion or discontinuation of adjuvant osimertinib.
5. Histologically/cytologically confirmed nonsquamous NSCLC (Investigators confirmed recurrence of primary lesion allowed if biopsy not available)
6. No prior systemic anti-cancer therapy after adjuvant therapy, but can receive local therapy (including surgery, radiotherapy, etc. per investigator choice).
7. Patients with asymptomatic or stable CNS metastases allowed.

Inclusion Criteria for screening:

1. Male or female, at least 18 years of age. Type of patient and disease characteristics
2. EGFR mutation (Exon 19del/Exon 21 L858R)-reconfirmed for study entry (mandatory undergo NGS by plasma, and tissue if applicable).
3. Life expectancy >12 weeks at Day 1.

Exclusion Criteria:

1. Patients with only local/regional recurrence.
2. Spinal cord compression and symptomatic brain metastases.
3. Past medical history of ILD, drug-induced ILD, radiation pneumonitis that required steroid treatment, or any evidence of clinically active ILD.
4. Adjuvant osimertinib therapy was discontinued due to the occurrence of severe adverse events.
5. Prior with other adjuvant EGFR-TKIs (excluding osimertinib).
6. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the formulated product or previous significant bowel resection that would preclude adequate absorption of osimertinib.
7. History of hypersensitivity to active or inactive excipients of osimertinib or drugs with a similar chemical structure or class to osimertinib.
8. Contraindication for pemetrexed and cisplatin/carboplatin according to local approved label.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2030-05-18 (Estimated); Study Completion 2030-05-18 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of osimertinib + chemotherapy by evaluation of PFS in patients who had distant recurrence after adjuvant osimertinib. | Approximately 52 months
  PFS is defined as the time from initiation of osimertinib combined with chemotherapy until progression per RECIST 1.1 as assessed by the investigator at local site, or death due to any cause.
  The analysis will include all patients who successfully enrolled in the study, satisfied all inclusion/exclusion criteria and have taken at least one dose of osimertinib plus chemotherapy. All events will be included, regardless of whether the patient withdraws from therapy, receives another anti-cancer therapy or clinically progresses prior to RECIST 1.1 progression. However, if the patient progresses or dies immediately after two or more consecutive missed visits, the patient will be censored at the time of the latest evaluable assessment prior to the two missed visits.
  The primary measure of interest is the median PFS.

SECONDARY OUTCOMES:
ORR | Approximately 52 months
  ORR is defined as the proportion of patients who have a confirmed CR or confirmed PR as determined by the investigator at local site per RECIST 1.1.
  The analysis will include all enrolled patients have taken at least one dose of osi plus chemotherapy. Data obtained from first dose up until progression, or the last evaluable assessment in the absence of progression will be included in the assessment of ORR, regardless of whether the patient withdraws from therapy. Patient who discontinues treatment without a response or progression, receive a subsequent therapy, and then respond will not be included as responder in the ORR.
TTD | Approximately 52 months
  TTD is defined as time from first dose of osimertinib + chemotherapy until discontinuation of treatment for any reason, including disease progression, toxicity, and death. The analysis will include all patients who successfully enrolled in the study, satisfied all inclusion/exclusion criteria and have taken at least one dose of osimertinib plus chemotherapy. Median TTD will be described.
depth of response | Approximately 52 months
  Depth of response (ie, tumour shrinkage/change in tumour size) by investigator assessment at local site was defined as the relative change in the sum of the longest diameters of RECIST target lesions at the nadir in the absence of new lesions or progression of non-target lesions compared to baseline.
DCR | Approximately 52 months
  DCR is defined as the percentage of patients who have a confirmed CR/PR or who have SD for at least 6 weeks minus 1 week per RECIST 1.1 as assessed by local site after date of first dose.
DoR | Approximately 52 months
  DoR is defined as the time from the date of first documented confirmed response until date of documented progression per RECIST 1.1 as assessed by the investigator at local site or death due to any cause.
  The primary measure of interest is the median DoR.
OS | Approximately 52 months
  OS is defined as time from first dose of osimertinib and chemotherapy until the date of death due to any cause.
  Landmark rate at 36 months of OS will be described.

OTHER OUTCOMES:
safety and tolerability | Approximately 52 months
  Safety and tolerability will be evaluated in terms of AEs (graded by CTCAE v5), vital signs (pulse and blood pressure), clinical laboratory, physical examination, ECG parameters, LVEF, and ECOG Performance Status.

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Kunming
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org.
  Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/